CLINICAL TRIAL: NCT02503423
Title: Phase 1-2 Study of the Safety, Pharmacokinetics, and Preliminary Activity of ASTX660 in Subjects With Advanced Solid Tumors and Lymphomas
Brief Title: Phase 1-2 Study of ASTX660 in Subjects With Advanced Solid Tumors and Lymphomas
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASTX660-01
Record Dates: First submitted 2015-07-02; First posted 2015-07-21 (Estimated); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumors; Lymphoma
Keywords: cervical cancer; HNSCC; CTCL; PTCL; DLBCL
MeSH Terms: conditions — Lymphoma; Uterine Cervical Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — ASTX-660

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Phase 1 - Part 1 (completed) (Experimental): Dose-escalation stage to identify the MTD and the RP2D, defined as either the MTD or a dose below the MTD that the Data and Safety Review Committee (DSRC) agree shows adequate pharmacological evidence of target engagement and/or clinical activity. Subjects will receive ASTX660 once a day for 7 consecutive days every other week of each 28-day cycle (ie, [7 days on/ 7 days off] ×2; daily dosing on Days 1-7 and 15-21). The starting dose will be escalated stepwise in successive cohorts of 3 to 6 evaluable subjects each (standard 3+3 study design), until the RP2D is determined.
  Interventions: Drug: ASTX660
- Phase 1 - Part 2 (completed) (Experimental): Dose-expansion stage to confirm tolerability of ASTX660 at the RP2D using the every-other-week daily dosing regimen. Up to a total of 12 subjects (including the 3 or 6 subjects treated at the RP2D in Part 1) will be treated at the RP2D.
  Interventions: Drug: ASTX660
- Phase 1 - Part 3 (optional) (Experimental): The purpose of the optional Part 3 is to allow for exploration of an alternative dosing regimen of ASTX660 based on emerging safety, PK, and pharmacodynamic (PD) data from Parts 1 and 2 (using the original every-other-week dosing regimen), with agreement of the DSRC. If Part 3 is conducted, the plan is to enroll up to 18 evaluable subjects in 1 or more cohorts using a standard 3+3 study design.
  Interventions: Drug: ASTX660
- Phase 2 - Cohort 1 (Experimental): Treatment with ASTX660 for recurrent/metastatic head and neck squamous cell carcinoma (HNSCC) not responsive or relapsed after standard therapy.
  Interventions: Drug: ASTX660
- Phase 2 - Cohort 2 (Experimental): Treatment with ASTX660 for relapsed or refractory diffuse large B-cell lymphoma (DLBCL).
  Interventions: Drug: ASTX660
- Phase 2 - Cohort 3 (Experimental): Treatment with ASTX660 for progressive or relapsed peripheral T-cell lymphoma (PTCL).
  Interventions: Drug: ASTX660
- Phase 2 - Cohort 4 (Experimental): Treatment with ASTX660 for relapsed or refractory cutaneous T-cell lymphoma (CTCL).
  Interventions: Drug: ASTX660
- Phase 2 - Cohort 5 (Experimental): Treatment with ASTX660 for other tumor types that are characterized by a molecular feature that may confer sensitivity to ASTX660 (eg, oncogenic activation of the NF-κB pathway or documented amplification of the gene loci encoding c-IAP1 or c-IAP2), pending confirmation in writing by the Astex medical monitor.
  Interventions: Drug: ASTX660
- Phase 2 - Cohort 6 (Experimental): Treatment with ASTX660 for cervical carcinoma not responsive or relapsed after standard therapy.
  Interventions: Drug: ASTX660

INTERVENTIONS:
Drug: ASTX660 — described above
  Other Names: Treatment of ASTX660 for advanced solid tumors and lymphomas

SUMMARY:
This is an open-label, dose-escalation Phase 1/2 study to assess the safety of ASTX660, determine the maximum tolerated dose (MTD), recommended Phase 2 dose (RP2D), and recommended dosing regimen, and to obtain preliminary efficacy, pharmacokinetic (PK), and target engagement data, in subjects with advanced solid tumors or lymphoma for whom standard life-prolonging measures are not available.

DETAILED DESCRIPTION:
ASTX660 is a synthetic small molecule dual antagonist of cellular inhibitor of apoptosis protein (cIAP) 1 and X-linked inhibitor of apoptosis protein (XIAP) that has been shown to have potent proapoptotic and tumor growth inhibitory activity in nonclinical models. The Phase 1 portion of the study (completed) will determine the MTD, RP2D, and recommended dosing regimen. The Phase 2 portion will evaluate activity in selected tumor types. Subjects will continue to receive their assigned treatment throughout the study until the occurrence of disease progression, death, or unacceptable treatment-related toxicity, or until the study is closed by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and comply with the protocol and study procedures, understand the risks involved in the study, and provide written informed consent before any study-specific procedure is performed.
2. Men and women 18 years of age or older.
3. Subjects with histologically or cytologically confirmed advanced solid tumors or lymphoma that is metastatic or unresectable, and for whom standard life-prolonging measures are not available. Specific tumor types that will be selected for study in Phase 2 are detailed in the protocol.

   a. For Phase 2 Cohort 3, subjects must have histologically confirmed PTCL (local pathology report) as defined by 2016 World Health Organization (WHO) classification. The following subtypes are eligible for the study: adult T-cell lymphoma/leukemia, extranodal natural killer (NK)/T-cell lymphoma nasal type, enteropathy-associated T-cell lymphoma, monomorphic epitheliotropic intestinal T-cell lymphoma, hepatosplenic T-cell lymphoma, subcutaneous panniculitis-like T-cell lymphoma, peripheral T-cell lymphoma not otherwise specified, angioimmunoblastic T-cell lymphoma, follicular T-cell lymphoma, nodal peripheral T-cell with T-follicular helper (THF) phenotype, and anaplastic large-cell lymphoma.
4. For Phase 2 Cohorts 3 and 4, patients must have evidence of documented progressive disease and must have received at least two prior systemic therapies.

   1. Subjects with CD30-positive lymphoma must have received, be ineligible for, or intolerant to brentuximab vedotin, provided that brentuximab vedotin is locally approved and available.
   2. Subjects with mycosis fungoides or Sezary syndrome must have received, be ineligible or intolerant to mogamulizumab, provided that mogamulizumab is locally approved and available.
5. In the Phase 2 portion of the protocol only, subjects must have measurable disease according to response criteria appropriate for their type of cancer.

   a. For Phase 2 Cohort 3 (PTCL), measurable disease by contrast-enhanced diagnostic CT (at least 1 nodal lesion >1.5 cm or extranodal lesions >1.0 cm) is required.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
7. Acceptable organ function, as evidenced by the following laboratory data:

   1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <=2.0 * upper limit of normal (ULN).
   2. Total serum bilirubin <=1.5 * ULN
   3. Absolute neutrophil count (ANC):

      * Phase 1 and 2 (except Phase 2 subjects with known lymphoma; ie, not applicable for Cohorts 3 or 4) >=1500 cells/mm3
      * Phase 2 subjects with known lymphoma: >=1000 cells/mm3 (>750 cell/mm3 for subjects with lymphoma in bone marrow)
   4. Platelet count:

      * Phase 1 and 2 (except Phase 2 subject with known lymphoma; ie, not applicable for Cohorts 3 or 4) >=100,000 cells/mm3
      * Phase 2 subjects with known lymphoma: >= 50,000 cells/mm3; >=25,000 cells/mm3 for subjects with lymphoma in bone marrow
   5. Serum creatinine levels <= 1.5 * ULN, or calculated (by Cockcroft-Gault formula or other accepted formula) or measure creatinine clearance >=50 mL/min.
   6. Amylase and lipase <=ULN.
8. Women of child-bearing potential (according to recommendations of the Clinical Trial Facilitation Group [CTFG]; see protocol for details) must not be pregnant or breastfeeding and must have a negative pregnancy test at screening. Women of child-bearing potential and men with female partners of child-bearing potential must agree to practice 2 highly effective contraceptive measures of birth control (as described in the protocol) and must agree not to become pregnant or father a child while receiving treatment with study drug and for at least 3 months after completing treatment. Contraceptive measures which may be considered highly effective comprise combined hormonal contraception (oral, vaginal, or transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, sexual abstinence, and surgically successful vasectomy. Abstinence is acceptable only if it is consistent with the preferred and usual lifestyle of the subject. Periodic abstinence (eg, calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of birth control.

Exclusion Criteria:

1. Hypersensitivity to ASTX660, excipients of the drug product, or other components of the study treatment regimen.
2. Poor medical risk because of systemic diseases (e.g. active uncontrolled infections) in addition to the qualifying disease under study.
3. Life-threatening illness, significant organ system dysfunction, or other condition that, in the investigator's opinion, could compromise subject safety or the integrity of the study outcomes, or interfere with the absorption or metabolism of ASTX660.
4. History of, or at risk for, cardiac disease, as evidenced by 1 or more of the following conditions:

   1. Abnormal left ventricular ejection fraction (LVEF; <50%) or echocardiogram ECHO or multiple gated acquisition scan (MUGA).
   2. Congestive cardiac failure of >= Grade 3 severity according to New York Heart Association (NYHA) functional classification defined as subjects with marked limitation of activity and who are comfortable only at rest.
   3. Unstable cardiac disease including angina or hypertension as defined by the need for overnight hospital admission within the last 3 months (90 days).
   4. History or presence of complete left bundle branch block, heart block, cardiac pacemaker or significant arrhythmia.
   5. Concurrent treatment with any medical that prolongs QT interval and may induce torsades de pointes, and which cannot be discontinued at least 2 weeks before treatment with ASTX660. [Applies to Phase 1 only].
   6. Personal history of long QTc syndrome or ventricular arrhythmias including ventricular bigeminy.
   7. Screening 12-lead ECG with measurable QTc interval (according to either Fridericia's or Bazett's correction) of >=470 msec).
   8. Any other condition that, in the opinion of the investigator, could put the subject at increased cardiac risk.
5. Known history of human immunodeficiency virus (HIV) infection, or seropositive results consistent with active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection.
6. Grade 2 or greater neuropathy [Applies to Phase 1]. Grade 3 or greater neuropathy [Applies to Phase 2].
7. Known brain metastases, unless stable or previously treated.
8. Known significant mental illness or other conditions such as active alcohol or other substance abuse that, in the opinion of the investigator, predisposes the subject to high risk of noncompliance with the protocol treatment or assessments.
9. Prior anticancer treatments or therapies within the indicated time window prior to first dose of study treatment (ASTX660), as follows:

   1. Cytotoxic chemotherapy or radiotherapy within 3 weeks prior and any encountered treatment-related toxicities (excepting alopecia) not resolved to Grade 1 or less [Phase 1] or Grade 2 or less [Phase 2].
   2. Skin directed treatments, including topicals and radiation within 2 weeks prior.
   3. Monoclonal antibodies within 4 weeks prior and any encountered treatment-related toxicities not resolved to Grade 1 or less [Phase 1] or Grade 2 or less [Phase 2].
   4. Small molecules or biologics (investigational or approved) within the longer of 2 weeks or 5 half-lives prior to study treatment and any encountered treatment-related toxicities not resolved to Grade 1 or less [Phase 1] or Grade 2 or less [Phase 2].
   5. At least 6 weeks must have elapsed since CAR-T infusion and subjects must have experienced disease progression, and not have residual circulating CAR-T cells in peripheral blood (based on local assessment). Any encountered treatment-related toxicities must have resolved to Grade ≤1.
10. Concurrent second malignancy currently requiring active therapy, except breast or prostate cancer stable on or responding to endocrine therapy or superficial bladder cancer [Phase 2].
11. Known central nervous system (CNS) lymphoma [Phase 2].
12. Patients with a history of allogenic transplant must not have ≥Grade 3 graft-versus-host disease (GVHD) or any clinically significant GVHD requiring systemic immunosuppression [Phase 2].
13. Systemic corticosteroids >20 mg prednisone equivalent (unless patient has been taking a continuous dose for >3 weeks prior to study entry and there is documented radiological progression) [Phase 2]. Stable dose of medium or low potency topical corticosteroids for at least 3 weeks prior to study entry are permitted [Phase 2].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety (Phase 1) - number of subjects with AEs, DLTs, abnormal clinical laboratory values or physical exam results | Up to 78 months
  Incidence of dose-limiting toxicities (DLTs) and other adverse events (AEs)
Efficacy (Phase 2) - antitumor activity assessed by objective response rate (ORR) | Up to 84 months
  Antitumor activity by objective response rate
Efficacy (Phase 2) - antitumor activity assessed by disease control rate (DCR) | Up to 84 months
  Antitumor activity by disease control rate

SECONDARY OUTCOMES:
Pharmacokinetic outcome of concentration-time curve (AUC) | First 9 weeks of study treatment
  Assessment of pharmacokinetic parameter area under the concentration-time curve (AUC).
Pharmacokinetic outcome of maximum concentration (Cmax) | First 9 weeks of study treatment
  Assessment of pharmacokinetic parameter maximum concentration (Cmax).
Pharmacokinetic outcome of minimum concentration (Cmin) | First 9 weeks of study treatment
  Assessment of pharmacokinetic parameter minimum concentration (Cmin).
Pharmacokinetic outcome of time to maximum concentration (Tmax) | First 9 weeks of study treatment
  Assessment of pharmacokinetic parameter time to maximum concentration (Tmax)
Pharmacokinetic outcome of samples over time | First 9 weeks of study treatment
  Assessment of pharmacokinetic parameter elimination half life (t½).
Pharmacokinetic outcome of samples over time | First 9 weeks of study treatment
  Assessment of pharmacokinetic parameter of other secondary PK parameters of ASTX660 if data permit.
Pharmacokinetic outcome of analysis of ASTX660 metabolites if applicable | First 9 weeks of study treatment
  Assessment of pharmacokinetic parameter analysis of ASTX660 metabolites if applicable.
Duration of antitumor response | Up to 84 months
  Time from the date of the earliest assessment of complete response or partial response to the date of relapse or death, whichever occurs earlier, or the last efficacy assessment date for subjects without a relapse or death.
Progression-free survival | Up to 84 months
  Number of days from the start of the study treatment to disease progression or death, whichever occurs first.
Overall survival | Up to 84 months
  Number of days from the day the subject received the first study treatment to the date of death, regardless of cause.
Assessment of target (cIAP1) engagement | Up to 84 months
  Percentage degradation of cIAP1 protein in PBMCs from baseline, in response to ASTX660 treatment.

CONTACTS AND LOCATIONS:
Locations (68):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - HonorHealth Research Institute, Scottsdale, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Simlow Cancer Hospital at Yale, New Haven, Connecticut
  - Emory University winship Cancer Institute, Atlanta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - The Sidney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Dartmouth-Hitchcock Medical Center (DHMC), Lebanon, New Hampshire
  - Summit Medical Group - Florham Park Campus/Atlantic Health, Florham Park, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York University Langone Medical Center, New York, New York
  - New York Presbyterian Hospital Columbia University Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Rochester Skin Lymphoma Medical Group, Rochester, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - The Ohio State University and Wexner Medical Center, James Cancer Hospital, Columbus, Ohio
  - University of Oklahoma Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Hollings Cancer Center, Charleston, South Carolina
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - CliniCore Texas, Houston, Texas
  - START- South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - Virgina Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle Cancer Care Alliance, Seattle, Washington
- Belgium (3):
  - Centre Hospitalier Universitaire Universite Catholique de Louvain - Site Godinne, Yvoir, Namur
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - Intitut Jules Boredt, Brussels
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Nova Scotia Health Athority-Qeii HSC, Halifax, Nova Scotia
  - Sunnybrook Hospital, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- France (7):
  - Gustave Roussy Cancer Campus (IGR), Villejuif, Cedex
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Lyon
  - Institut Bergonié, Unicancer, Bordeaux
  - Centre Antoine Lacassagne, Oncologie Médicale, Nice
  - Centre Henri Becquerel, Hematology, Rouen
  - Institut Universitaire du Cancer - Oncopôle, Department d'Hématologie, Toulouse
  - CRU de Tours - Hôpital Bretonneau, Hématologie -Thérapy Cellulaire, Tours
- Hungary (3):
  - Semmelweis Egyetem - I. sz. Belgyógyászati Klinika, Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Szabolcs-Szatmár-Bereg Megyei Kórházak És Egyetemi Oktatókórház, Nyíregyháza
- Italy (4):
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico Sant Orsola-Malpighi, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - Instituto Europeo di Oncologia, Milan
  - Azienda Socio Santaria Territoriale Monza- Osperdale San Gerado, Monza
- Spain (4):
  - Institut Catala d'Oncologia, Girona, Giona
  - imCORE - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Fundacion Jimenez Diaz Preview, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (9):
  - University Hospitals of Leicester NHS Trust, Leicester, East Midlands
  - University Hospital Southhampton NHS Foundation Trust - Somers Cancer Research, Southampton, Hampshire
  - Churchill Hospital, Oxford University Hospital NHS Trust, Oxford, Oxfordshire
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital, Birmingham
  - Beatson Cancer Center and University of Glasgow, Glasgow
  - University College London Hospitals NHS Foundation Trust, London
  - Guy's and Saint Thomas' NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Christie Hospital, Manchester

REFERENCES:
- [Derived] Johnson CN, Ahn JS, Buck IM, Chiarparin E, Day JEH, Hopkins A, Howard S, Lewis EJ, Martins V, Millemaggi A, Munck JM, Page LW, Peakman T, Reader M, Rich SJ, Saxty G, Smyth T, Thompson NT, Ward GA, Williams PA, Wilsher NE, Chessari G. A Fragment-Derived Clinical Candidate for Antagonism of X-Linked and Cellular Inhibitor of Apoptosis Proteins: 1-(6-[(4-Fluorophenyl)methyl]-5-(hydroxymethyl)-3,3-dimethyl-1 H,2 H,3 H-pyrrolo[3,2- b]pyridin-1-yl)-2-[(2 R,5 R)-5-methyl-2-([(3R)-3-methylmorpholin-4-yl]methyl)piperazin-1-yl]ethan-1-one (ASTX660). J Med Chem. 2018 Aug 23;61(16):7314-7329. doi: 10.1021/acs.jmedchem.8b00900. Epub 2018 Aug 9. PMID 30091600